CLINICAL TRIAL: NCT06281860
Title: Phase I Clinical Trial Testing the Dose Escalation and Expansion of Pressurized IntraThoracic Hyperthermic Aerosol Cisplatin Administration for the Management of Pleural Carcinosis
Brief Title: Treatment Pleural Carcinosis of Pressurized IntraThoracic Hyperthermic Aerosol Cisplatin Administration
Acronym: PITHAC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dr Jean Yannis PERENTES (Other)
Responsible Party: Sponsor-Investigator, Dr Jean Yannis PERENTES, Sponsor-Investigator, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PITHAC; 2023-00099 (Registry Identifier: BASEC)
Record Dates: First submitted 2023-09-16; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung; Carcinoma Breast Stage IV; Ovarian Cancer; Esophageal Cancer; Gastric Cancer
Keywords: Pressurized intrathoracic hyperthermic aerosol chemotherapy
MeSH Terms: conditions — Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Ovarian Neoplasms; Esophageal Neoplasms; Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomised monocentric Phase I clinical trial study with cisplatin dose escalation administered by PITHAC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohorte 1 _ 7.5 mg/m2 (Experimental): cohorte 1: 7.5 mg/m2 of cisplatin (once)
  Interventions: Drug: Cisplatine Teva®
- Cohorte 2 _ 12.5 mg/m2 (Experimental): cohorte 2: 12.5 mg/m2 of cisplatin (once)
  Interventions: Drug: Cisplatine Teva®
- cohorte 3: 35 mg/m2 of cisplatin (Experimental): cohorte 3: 35 mg/m2 of cisplatin (once)
  Interventions: Drug: Cisplatine Teva®
- cohorte 4: 70 mg/m2 of cisplatin (Experimental): cohorte 4: 70 mg/m2 of cisplatin (once)
  Interventions: Drug: Cisplatine Teva®

INTERVENTIONS:
Drug: Cisplatine Teva® — PITHAC: Cisplatin (Cisplatine Teva®) at a dose between 7.5 and 70 mg/m2 of body surface at a temperature of 39±1°C
  Other Names: Procedure/Surgery

SUMMARY:
Within the context of pleural carcinosis, the present study is a dose escalation with determination of the maximum tolerated doses (MTD) of pressurized cisplatin administration associated to moderate hyperthermia in the pleura. This will be followed by an expansion phase at the recommended dose (RD).

DETAILED DESCRIPTION:
Adverse events: the evaluation of the safety of cisplatin administered by PITHAC is the primary endpoint of both parts of the study Cisplatin administration will be performed on D0. Postoperative pain management according to the Enhanced Recovery After Surgery program following the surgical procedure.

Dyspnoea score will be scored at screening, and every day until D10 and checked one last time at D30 using the CR-10 scale.

Chest X-ray will be performed at screening, D0, 24h post intervention, D10 and D30.

Monitoring of adverse events (AEs), serious and non-serious, will be conducted throughout the study from the surgery.

Blood samples for cisplatin pharmacokinetics PK will be performed on D0 pre-intervention, 12h post intervention, 24h and 48h post intervention.

Translational blood tests for immune profiling will be performed on D0 pre-intervention, D10 and D30. Translational blood tests on inflammatory cytokine assessment will be performed on D0 pre-intervention, 12h post intervention, 24h, 48h and on D10 and D30. Tissue biopsy for free cisplatin PK and Pleural biopsy for tissue immune infiltration will be performed on D0 before and after treatment administration.

Malignant pleural effusion (MPE) assessment: Immune environment and neoantigen landscape will be collected before the PITHAC procedure and via the indwelling pleural catheter (D0, at hospital discharge and D10).

STATISTICAL METHODS:

PART A: Dose escalation and MTD determination: The sample size is set to determine the MTD by using the 3+3 design. Cohorts of 3-6 patients will be recruited sequentially at each of the cisplatin doses. The total number of patients is expected to be 12 with a maximum of 24, depending on the level of MTD. If there are patients who are not evaluable for the objectives in the study, additional patients will be enrolled. Patients not evaluable will be replaced but not withdrawal from the study.

Primary Analysis: dose limiting toxicities; To determine the maximum tolerated dose (MTD) of cisplatin administered with PITHAC, the primary study outcome is the occurrence of Dose Limiting Toxicities (DLT). The number and proportion of patients with DLTs will be presented overall and by dose and will be plotted vs dose. The MTD will be graphically displayed. Secondary Analyses: safety profile of cisplatin administered with PITHAC: The safety analysis will be performed on the safety population. -Treatment emergent AE frequencies will be summarised by system organ class and preferred term (MedDRA) overall and by dose. AEs will also be tabulated by system organ class and preferred term including maximum severity grade according to the NCI-CTCAE criteria version 5 and relationship to treatment. Incidence of treatment discontinuations due to AEs and SAEs will be summarised overall and by dose. -Safety Lab parameters and vital signs at pre-treatment and post-treatment and corresponding changes from pre-treatment will be presented by dose as descriptive statistics. Efficacy analysis will be performed on efficacy population. Dyspnoea will be scored from screening to D30. Dyspnoea score will be presented at pre- and post-treatment and change from pre- to post-treatment will be presented as descriptive statistics by dose. The pleural infusion index will be determined by comparing chest X-rays before treatment (D0) and post-treatment at D1, D10 and 30 days and pleurodesis or indwelling catheter placement. The index will be presented at pre- and post-treatment and change from pre- to post-treatment will be presented as descriptive statistics by dose. Exploratory endpoints: exploratory analyses will be performed by tissue immunostaining and image analysis will be carried out. The concentration of cisplatin in tumor tissue at the beginning and end of mild hyperthermia PITHAC will be evaluated by Laser Ablation Inductively Coupled Plasma Mass Spectrometry (LA-ICP-MS) that will allow visualization of cisplatin distribution and penetration in tumor biopsies. The correlation between cisplatin concentration and penetration into tumor tissue and clinical response will be explored. Immune infiltration in tumor tissues will be assessed by immunostainings and image analysis will be performed. Immune cells proportions in peripheral blood before and after PITHAC at D0, 10 and 30 will be explored using DURAClone Panels for flow cytometry.

PART B: Expansion: Determination of Sample Size: the sample in the expansion phase is not based on a formal hypothesis. To evaluate the safety of cisplatin administered by PITHAC at the RD and undertake an initial evaluation of efficacy, a total of 15 patients will be enrolled in this exploratory part of the study. Statistical criteria of termination of trial: there are no statistical criteria of termination of the trial in this part of the study.

Primary Analysis: dose limiting toxicities; To determine the maximum tolerated dose (MTD) of cisplatin administered with PITHAC, the primary study outcome is the occurrence of Dose Limiting Toxicities (DLT). The number and proportion of patients with DLTs will be presented overall and by dose and will be plotted vs dose. The MTD will be graphically displayed. Secondary Analyses: safety profile of cisplatin administered with PITHAC: The safety analysis will be performed on the safety population. -Treatment emergent AE frequencies will be summarised by system organ class and preferred term (MedDRA) overall and by dose. AEs will also be tabulated by system organ class and preferred term including maximum severity grade according to the NCI-CTCAE criteria version 5 and relationship to treatment. Incidence of treatment discontinuations due to AEs and SAEs will be summarised overall and by dose. -Safety Lab parameters and vital signs at pre-treatment and post-treatment and corresponding changes from pre-treatment will be presented by dose as descriptive statistics. Efficacy analysis will be performed on efficacy population. Dyspnoea will be scored from screening to D30. Dyspnoea score will be presented at pre- and post-treatment and change from pre- to post-treatment will be presented as descriptive statistics by dose. The pleural infusion index will be determined by comparing chest X-rays before treatment (D0) and post-treatment at D1, D10 and 30 days and pleurodesis or indwelling catheter placement. The index will be presented at pre- and post-treatment and change from pre- to post-treatment will be presented as descriptive statistics by dose. Exploratory endpoints: exploratory analyses will be performed by tissue immunostaining and image analysis will be carried out. The concentration of cisplatin in tumor tissue at the beginning and end of mild hyperthermia PITHAC will be evaluated by Laser Ablation Inductively Coupled Plasma Mass Spectrometry (LA-ICP-MS) that will allow visualization of cisplatin distribution and penetration in tumor biopsies. The correlation between cisplatin concentration and penetration into tumor tissue and clinical response will be explored. Immune infiltration in tumor tissues will be assessed by immunostainings and image analysis will be performed. Immune cells proportions in peripheral blood before and after PITHAC at D0, 10 and 30 will be explored using DURAClone Panels for flow cytometry.

QUALITY ASSURANCE AND CONTROL: all data collected will be coded and recorded on the RedCap search software. The conformity of eCRF with protocol specifications is checked and validated by the SI and/or qualified individuals, according to ICH GCP. Case Report Forms (eCRF): electronic data entry will be performed via a web-based application (REDCap). Security passwords will be provided to each properly trained investigator. An eCRF for data collection will be developed in Redcap. The REDCap database will record the data obtained with the coding number specific to each patient: this code will consist of PITHAC-01, PITHAC-02 etc…. A specific subject identification log will be compiled to record the identifying information of enrolled participants, providing the link to individual attributed codes. This document (word file) will be kept separately, it will be password protected and saved in a secure directory on a CHUV server. At the end of the project, the subject identification log will be kept by the principal investigator. Best practices will be adopted to ensure that data are complete, reliable, and processed correctly, thus providing high-quality data, keeping the number of errors and missing data as low as possible, and gathering a maximum amount of accurate data for analysis. The data collected through RedCap® will be automatically checked by the implementation of data validation rules (e.g., data-type, maximum/minimum range, missing data checks, and other logical tests) and automatic alerts. Specification of source documents: study monitors will perform ongoing source data verification to confirm that critical protocol data (i.e., source data) entered into the eCRFs by authorized site personnel are accurate, complete, and verifiable from source documents. Source documents (paper or electronic) are those in which patient data are recorded and documented for the first time. They include, but are not limited to, hospital records, clinical and office charts, laboratory notes, memoranda, evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies of transcriptions that are certified after verification as being accurate and complete, X-rays, patient files, and records kept at pharmacies, laboratories, and medico-technical departments involved in the clinical trial. The Investigator must keep a subject file (medical file, original medical records) electronically (SOARIAN/ARCHIMEDE) for every subject included in the trial. All documents containing source data must be filed in the electronic patient file. Electronic subject files (SOARIAN/ARCHIMEDE) will be accessible to the Monitor to perform source data verification. Record keeping / archiving: the SI will retain copies of the patient trial records (CRFs, patient informed consent statement, drug inventory logs and all other information collected during the trial) and documentation until at least 10 years after the termination of the trial.It must be available for review by the Monitor and must be ready for Sponsor audit as well as for inspection by Competent Authorities during and after the trial and must be safely archived for at least 10 years (or per local requirements or as otherwise notified by the Sponsor) after the end of the trial. The documents to be thus archived include the Subject Identification List and the signed subject ICFs.

Safety Monitoring (Dose Escalation Part): a Trial Safety Board (TSB) will be constituted for the part A of the trial, being responsible for maintaining the scientific integrity of the trial and safety of patients. This Board will review the DLTs of each cohort and decide whether to escalate or not to the next dose level (next cohort). Details on the dose escalation design, rules, and the role of the TSB are provided in the DEP. The TSB will give the green light to start part B after recommended dose confirmation, based on safety and efficacy data of all patients enrolled in part A. For Part B, the responsibility for the safety of the individual patient lies with the investigator and the SI. Clinical Trial Monitoring: clinical monitoring activities have the ultimate purpose to guarantee that the rights and well-being of human subjects are protected, that the reported study data are accurate, complete and verifiable from source documents, and that the conduct of the study complies with the latest approved version of the study protocol, with ICH-GCP guidelines and applicable regulations .

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Body weight at least 30 kg
* Eastern cooperative oncology group performance status score of 0-2 at enrolment
* Patient with pleural carcinosis that qualify for a surgical intervention for pleurodesis or placement of an indwelling permanent catheter.
* Life expectancy of at least 3 months
* Pathology-confirmed pleural carcinosis with malignant pleural effusion (either histological confirmation is already available based on a previous tru-cut pleural biopsy or previous pleural fluid cytology is positive for malignant cells or high suspicion of pleural carcinosis based on computed tomography imaging which must be confirmed by fresh frozen section analyses of tissue harvested during pithac operative procedure)
* Non-small cell lung cancer, breast cancer, lymphoma, ovarian cancer, oesophageal cancer, gastric cancer, and malignant tumour of the serous membranes (mesothelioma) confirmed by pathology either as part of a diagnostic workup of suspected pleural carcinosis OR available from other previous examinations patients undergoing a planned videothoracoscopy to perform pleurodesis or a placement of a tunnelled catheter
* Adequate liver, kidney, and bone marrow functions as assessed by laboratory tests (serum total bilirubin <1.5 mg/dl, aspartate transaminase and alanine transaminase less than 2.5 times the upper limit of the normal range, creatinine clearance ≥60 ml/min, absolute neutrophil count ≥1,500/μl, haemoglobin ≥90 g/L, platelets ≥100,000/μl)
* I) Patients with past/resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible, if HBV DNA test is negative. Ii) HBV DNA must be obtained in patients with positive hepatitis B core antibody prior start of study treatment.
* Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA
* Adequate cardiac functions as assessed by echocardiography
* Adequate birth control measures
* Signed informed consent

Exclusion Criteria:

* Patients with active or chronic hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at pre-screening)
* Patients with active hepatitis C
* Any known formal contra-indication for video-assisted thoracoscopy (VATS) according to pulmonary and cardiac preliminary investigations.
* Systemic cytotoxic anticancer treatment within 10 days before and after enrolment except for inhibitors of vascular endothelial growth factor for which this period should be decided according to the used drug (for bevacizumab the period involves 4 weeks before and after enrolment, for lenvatinib 1 week before and 2 weeks after, and for sorafenib 1 week before and after), no limitations applied for immune checkpoint inhibitors
* Major surgery within 28 days prior to enrolment
* Any unresolved toxicity from previous anticancer therapy of grade ≥2 according to the CTCAE except for alopecia, vitiligo, and laboratory values considered as adequate in the inclusion criteria and any irreversible toxicity that is expected to have impact on the study results or be a contraindication for the planned surgical intervention or be worsened by the investigational procedure
* Long lasting exposure to corticosteroids
* Known allergy to platinum compounds
* Non-small cell lung cancer with egfr or alk mutations unless refractory to tyrosine kinase inhibitor (thus off treatment)
* Uncontrolled intercurrent illness
* Clinically relevant hearing loss or tinnitus
* Clinically relevant neuropathy
* Life-threatening conditions (uncontrolled systemic infection etc.)
* Previous administration (by any route) of a total cumulative dose of more than 500 mg/m2 of cisplatin
* Secondary resistance to platinum compounds defined as tumour progression during platinum treatment or within 6 months after its cessation
* pregnancy
* judgement of the investigator that the patient is unlikely to comply with the study requirements
* current enrolment in another prospective clinical trial
* Incapacity of judgement
* Patients in emergency situation
* Myelossupression
* Yellow fever vaccine
* Concurrent prophylactic use of phenytoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 39 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation and Maximum Tolerated Dose determination (Part A): | 18 months approximately
  In order to determine the maximum tolerated dose (MTD) of cisplatin administered by PITHAC, the primary study outcome will be the occurrence of Dose Limiting Toxicities (DLT).
Expansion phase (Part B): | between 10 and 12 months
  Safety profile of cisplatin administered by PITHAC will be assessed by the incidence of Adverse Events and Serious Adverse Events according to NCI-CTCAE criteria (v5). Incidence and severity of intraoperative and post-operative complications will be measured using the Clavien-Dindo classification up to 30 days after the intervention.
  Safety profile of cisplatin administered by PITHAC will be assessed by the incidence of Adverse Events and Serious Adverse Events according to NCI-CTCAE criteria (v5). Incidence and severity of intraoperative and post-operative complications will be measured using the Clavien-Dindo classification up to 30 days after the intervention.

SECONDARY OUTCOMES:
Dose Escalation and MTD determination (Part A): | 18 months
  Safety profile of cisplatin administered with moderate hyperthermic PITHAC will be assessed by the incidence of Adverse Events and Serious Adverse Events according to NCI-CTCAE criteria (v5).
  Dyspnoea will be scored every day until Day 10 and re-evaluated at Day 30 after the procedure
  The pleural effusion index will be determined by comparing chest X-rays before, 24 hours (Day 0), at Day 10 and at Day 30 after PITHAC and pleurodesis or indwelling catheter placement
Expansion phase (Part B): | 10 /12 months
  Dyspnoea will be scored every day until Day 10 and re-evaluated at Day 30 after the procedure.
  The pleural effusion index will be determined by comparing chest X-rays before PITHAC procedure, 24 hours after, at Day 10 and Day 30 after PITHAC and pleurodesis or indwelling catheter placement.

OTHER OUTCOMES:
Dose Escalation and MTD determination (Part A):Exploratory outcomes | 18 months approximately
  Tissue immune infiltration will be assessed by comparing penetration depth and resulting immune infiltrate in pleural biopsy specimens at the beginning and at the end of PITHAC.
  The correlation between plasma concentrations of administered intrapleural cisplatin by PITHAC and acute secondary side effects will be evaluated.
  Tissue distribution of free cisplatin will be compared in pleural biopsy specimens at the beginning and at the end of PITHAC by gaz phase chromatography.
  Correlation between treatment outcome, percentage of cancer cell death, cisplatin concentration in pleural biopsies, release of pro-inflammatory proteins and the activation status of effector T-cell will be assessed.
  Assess the immune environment and immune responses mediated by neoantigen directed cytotoxic T cells (neoantigen landscape) in patient malignant pleural effusion (MPE) before and after PITHAC ((D0, 72h post intervention, Day 10 and D30).
Expansion phase (Part B):Exploratory outcomes | between 10 and 12 months
  Tissue immune infiltration will be assessed by comparing penetration depth and resulting immune infiltrate in pleural biopsy specimens at the beginning and at the end of PITHAC.
  The correlation between plasma concentrations of administered intrapleural cisplatin by PITHAC and acute secondary side effects will be evaluated.
  Tissue distribution of free cisplatin will be compared in pleural biopsy specimens at the beginning and at the end of PITHAC by gaz phase chromatography.
  Correlation between treatment outcome, percentage of cancer cell death, cisplatin concentration in pleural biopsies, release of pro-inflammatory proteins and the activation status of effector T-cell will be assessed.
  Assess the immune environment and immune responses mediated by neoantigen directed cytotoxic T cells (neoantigen landscape) in patient malignant pleural effusion (MPE) before and after PITHAC ((D0, 72h post intervention, Day 10 and D30).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yannis Perentes, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Chriqui LE, Abdelnour-Berchtold E, Zanfrini E, Devesa-Perez S, Gonzalez M, Krueger T, Ellefsen K, Destaillats A, Bonnet D, Hubner M, Bouchaab H, Bassani-Sternberg M, Peters S, Cavin S, Perentes JY. Phase I clinical trial testing the dose escalation and expansion of Pressurized IntraThoracic Hyperthermic Aerosol Cisplatin administration (PITHAC) for the management of pleural carcinosis. Cancer Treat Res Commun. 2024;42:100858. doi: 10.1016/j.ctarc.2024.100858. Epub 2024 Dec 17. PMID 39708537